CLINICAL TRIAL: NCT07177248
Title: Effects of a 12-Week Multicomponent Intervention on 24-Hour Movement Behaviour and Physical Fitness in Parents and Their Children: A Mediation Analysis
Brief Title: 12-Week Family-Based Multicomponent Program to Improve 24-Hour Movement Behaviors in Parents and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Valparaiso (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACTIBESE/FONDECYT 2023/1230801
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity; Sedentary Behaviors; Exercise; Sleep; Physical Fitness; Health Promotion
Keywords: Physical Activity; Sedentary Behavior; Sleep
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Non-randomized, two-arm, parallel study conducted in Chilean primary schools. Parent-child dyads were assigned by school-level scheduling/feasibility to either the multicomponent family-based program or usual activities. The intervention combined weekly digital guidance for parents and three family in-person sessions led by a Physical Education teacher. Outcomes were assessed at baseline and post-intervention (~Week 16). Analyses compare change scores between groups, adjusting for baseline and design features appropriate to non-randomized allocation.
Masking Description: Not applicable for this behavioral program; participants and providers were aware of group assignment. Standardized instructions and prespecified analyses were used to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Family-Based Multicomponent Program (Experimental): 12-week family-based program combining weekly parent digital guidance (infographics/videos + actionable tips) and three 90-min family sessions (functional training, modified games, outdoor trekking) led by a Physical Education teacher.
  Interventions: Behavioral: Family-Based 12-Week Multicomponent Program
- No Intervention: Usual Activities (No Intervention): Participants continue usual routines; same assessment schedule as the experimental arm.

INTERVENTIONS:
Behavioral: Family-Based 12-Week Multicomponent Program — Weekly digital materials to parents (email/WhatsApp) + three on-site sessions (~90 min each: functional training; modified games; outdoor trekking); 12 weeks total; delivered by a Physical Education teacher; attendance and delivery logs for fidelity.
  Other Names: Family Physical Activity Program
  Arms: Experimental: Family-Based Multicomponent Program

SUMMARY:
This study assessed a 12-week, family-oriented program intended to promote healthier 24-hour movement patterns among school-age children and their parents in Chile. Parent-child pairs volunteered from two private schools and one public school, and schools were used to determine group assignment in a parallel, non-randomized, open-label design.

The intervention blended brief weekly digital guidance for parents (concise infographics/videos and actionable tips sent via email/WhatsApp) with three in-person family sessions (a functional-training class, parent-child modified games, and an outdoor trekking activity) led by a Physical Education teacher with support from school staff. The comparison group continued usual routines and completed the same assessments.

Outcomes were collected at baseline and after the intervention period (post-intervention window around Week 16). The primary outcome was the change in children's out-of-school moderate-to-vigorous physical activity (MVPA) estimated with the Youth Activity Profile-Spain/Latin America version (YAP-SL). Secondary outcomes encompassed children's in-school and weekend MVPA, sedentary time, and sleep duration, as well as parents' MVPA and sedentary time (IPAQ-Short Form) and perceived physical fitness for both parents and children (International Fitness Scale, IFIS). Potential intervention-related adverse events during face-to-face activities and those reported between sessions were monitored.

The institutional ethics committee approved the protocol and the intervention was considered minimal risk. This is a retrospective registration completed after study execution at the request of the sponsor. An exploratory mediation analysis is planned to examine plausible pathways linking the program to changes in MVPA.

DETAILED DESCRIPTION:
Rationale Low physical activity and prolonged sedentary time in childhood are widespread and linked to unfavorable health and developmental outcomes. Engaging parents as agents of change is a promising strategy to support children's daily movement behaviors across the full 24-hour cycle (physical activity, sedentary time, and sleep). In Latin American school settings, pragmatic, scalable formats that combine short digital prompts with occasional on-site family activities may be feasible and impactful.

Objectives

1. Primary: Determine whether a 12-week multicomponent, family-based program increases children's out-of-school MVPA compared with usual activities.
2. Secondary: Evaluate effects on children's in-school and weekend MVPA, sedentary time, and sleep; parents' MVPA and sedentary time; and perceived physical fitness (parents and children).
3. Exploratory: Conduct a mediation analysis to explore potential pathways (e.g., changes in sedentary time, sleep, or perceived fitness) through which the intervention may influence children's MVPA.

Design and Setting Two-arm, parallel, non-randomized, open-label study conducted in Chilean primary schools. Group assignment was determined at the school level for logistical and feasibility reasons (two private and one public school). Assessments were completed at baseline and post-intervention (~Week 16).

Participants Eligible units were parent-child pairs recruited through school meetings. Children were primarily 5th-grade students (one school deviated for scheduling reasons). Inclusion required the ability to participate safely in light-to-moderate physical activity and access to email and/or WhatsApp for digital communications. Informed consent (parents) and assent (children) were obtained. Exclusions included medical conditions that would preclude safe participation or concurrent enrollment in another structured physical activity program.

Intervention (summary aligned with TIDieR)

* Format & Dose: 12 weeks combining weekly digital materials for parents and three on-site family sessions.
* Digital component (Weeks 4-15): Short infographics/videos and practical suggestions were delivered via email/WhatsApp each week (brief educational content early in the week and follow-up prompts later in the week).
* In-person sessions: (i) Functional training class for parents and children (school gym), (ii) modified games session (school gym), and (iii) outdoor trekking activity. Each lasted ~90 minutes and was supervised by a Physical Education teacher with assistance from the school's sports department.
* Implementation timeline (abridged): Week 1 school authorization; Week 2 information sessions and consent/assent; Week 3 baseline questionnaires and anthropometry; Weeks 4-15 digital materials; Weeks 7, 11, and 15 in-person sessions; Week 16 post-test; Week 17 feedback meetings with families and school authorities.
* Adherence & Fidelity: Delivery logs for digital materials and attendance records for on-site sessions were maintained; activities were adapted to accommodate varied fitness levels.

Comparator Participants in the comparison group maintained their usual activities and were measured on the same schedule as the intervention group.

Outcomes and Measurements

* Primary outcome: Children's out-of-school MVPA (min/day) estimated with the YAP-SL, which uses context-specific items and established calibration procedures to model daily MVPA.
* Secondary outcomes: Children's in-school and weekend MVPA (YAP-SL); sedentary time (hours/day, YAP-SL); sleep duration computed from weekday/weekend bed/wake times (average across the week); parents' MVPA and sedentary time derived from the IPAQ-Short Form; and perceived physical fitness for both parents and children using the International Fitness Scale (IFIS) (higher scores reflect better perceived fitness).
* Safety monitoring: Any intervention-related adverse events (e.g., musculoskeletal complaints, dizziness, falls) were recorded during face-to-face sessions and via parent reports between sessions.

Statistical Approach Primary analyses compare change from baseline to post-intervention between groups, with models adjusted for baseline values and additional covariates as appropriate for the non-randomized design. The mediation analysis will estimate indirect effects along pre-specified behavioral/fitness pathways using established regression-based procedures, recognizing design constraints and measured covariates.

Ethics and Oversight The study received approval from the institutional bioethics committee and adhered to the principles of the Declaration of Helsinki. Given the behavioral nature and low risk of the activities, monitoring was conducted by the research team, with procedures specified for reporting serious events to the PI and the ethics board.

Registration Note This is a retrospective registration finalized after data collection at the sponsor's request.

ELIGIBILITY:
Inclusion Criteria:

* Parent-child dyad from a participating primary school (child typically in grades 3-6).
* Parent/legal guardian aged ≥18 years; child aged ≥8 years at enrollment.
* Able to take part safely in light-to-moderate physical activity (medical clearance as needed).
* Access to a mobile phone with WhatsApp and/or email for weekly digital materials.
* Signed informed consent from the parent/legal guardian and assent from the child.
* Availability to attend the three scheduled in-person family sessions and complete baseline and post-intervention assessments.

Exclusion Criteria:

* Any medical condition, injury, or disability that, in the investigator's judgment, would make participation unsafe or preclude planned activities.
* Current participation in another structured physical activity or lifestyle intervention trial.
* Inability to comply with the study schedule, procedures, or outcome assessments.
* Lack of access to WhatsApp/email for receiving digital materials.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in children's out-of-school moderate-to-vigorous physical activity (MVPA), min/day | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  Daily minutes of MVPA estimated from the Youth Activity Profile-Spain/Latin America version (YAP-SL), using its established calibration procedure to convert item responses into minutes/day; higher values indicate more MVPA.

SECONDARY OUTCOMES:
Change in children's in-school MVPA, min/day | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  Minutes/day of MVPA during school time estimated with YAP-SL calibration; higher = more MVPA.
Change in children's weekend MVPA, min/day | (Weeks 1-3) and Post-intervention (~Week 16)
  Minutes/day of MVPA on weekend days derived from YAP-SL; higher = more MVPA.
Change in children's sedentary time, hours/day | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  Average daily sedentary time estimated from YAP-SL items; values expressed in hours/day; lower values indicate less sedentary behavior.
Change in children's sleep duration, hours/day | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  Sleep hours computed from reported bed- and wake-times for weekdays and weekends; weekly average calculated as (weekdayhours×5+weekendhours×2)/7; higher values indicate longer sleep duration.
Change in parents' MVPA, min/week | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  Weekly minutes of MVPA derived from the IPAQ-Short Form, computed as the sum of moderate + vigorous minutes/week in bouts ≥10 min. Per the IPAQ-SF scoring protocol, minutes at each intensity are truncated at 180 min/day to limit outliers; range 0-2 520 min/week; higher values indicate more MVPA.
Change in parents' sedentary time, hours/day | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  Average daily sitting time from the International Physical Activity Questionnaire-Short Form (IPAQ-SF), Sitting item. Reported for a usual weekday and expressed as hours/day; range 0-16 hours/day (equivalently 0-960 min/day). Higher values indicate more sedentary time.
Change in perceived physical fitness (parents and children), IFIS score (1-5) | Baseline (Weeks 1-3) and Post-intervention (~Week 16)
  International Fitness Scale (IFIS); five domains rated 1-5. Scores are averaged to obtain a domain-specific perceived fitness score; higher values reflect better perceived fitness.
Participants with intervention-related adverse events | Through study completion (up to 16 weeks).
  Count of participants reporting events plausibly related to the program during supervised sessions or between sessions (e.g., musculoskeletal complaints, dizziness, falls); events captured in session logs and via parent reports.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Javier Rodríguez-Rodríguez, PhD, Principal Investigator — Pontificia Universidad Católica de Valparaíso (PUCV)
Locations (1):
- Pontificia Universidad Católica de Valparaíso - School of Physical Education, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the main results will be shared, including parent-child demographics, group assignment, baseline and post-intervention outcomes (YAP-SL MVPA components, sedentary time, sleep measures), IPAQ-Short Form metrics, International Fitness Scale (IFIS) scores, and adverse event dataset. Direct identifiers will be removed; quasi-identifiers will be generalized (e.g., age in years; site masked). A data dictionary/codebook will accompany the dataset. Requests must be consistent with consent and ethics approvals.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after the Primary Completion Date and available for 36 months thereafter (extensions considered upon reasonable request).
Access Criteria: Available to qualified researchers with IRB/ethics approval and a signed Data Use Agreement. Requests should include a brief proposal and analysis plan and be sent to the Principal Investigator. Approved requests will receive access via a secure file transfer or institutional repository. Re-identification attempts and contact with participants/schools are prohibited; citation of the original study is required.

REFERENCES:
- [Background] Guagliano JM, Armitage SM, Brown HE, Coombes E, Fusco F, Hughes C, Jones AP, Morton KL, van Sluijs EMF. A whole family-based physical activity promotion intervention: findings from the families reporting every step to health (FRESH) pilot randomised controlled trial. Int J Behav Nutr Phys Act. 2020 Sep 22;17(1):120. doi: 10.1186/s12966-020-01025-3. PMID 32962724
- [Background] Hayes AF. Introduction to Mediation, Moderation, and Conditional Process Analysis: A Regression-Based Approach. 2nd ed. New York: Guilford Press; 2017.
- [Background] Zhao X, Lynch JG, Chen Q. Reconsidering Baron and Kenny: Myths and truths about mediation analysis. J Consum Res. 2010;37(2):197-206. https://doi.org/10.1086/651257
- [Background] Ortega FB, Ruiz JR, Espana-Romero V, Vicente-Rodriguez G, Martinez-Gomez D, Manios Y, Beghin L, Molnar D, Widhalm K, Moreno LA, Sjostrom M, Castillo MJ; HELENA study group. The International Fitness Scale (IFIS): usefulness of self-reported fitness in youth. Int J Epidemiol. 2011 Jun;40(3):701-11. doi: 10.1093/ije/dyr039. Epub 2011 Mar 24. PMID 21441238
- [Background] Fairclough SJ, Christian DL, Saint-Maurice PF, Hibbing PR, Noonan RJ, Welk GJ, Dixon PM, Boddy LM. Calibration and Validation of the Youth Activity Profile as a Physical Activity and Sedentary Behaviour Surveillance Tool for English Youth. Int J Environ Res Public Health. 2019 Oct 2;16(19):3711. doi: 10.3390/ijerph16193711. PMID 31581617
- [Background] Brand C, Zurita-Corvalan N, Batista Lemes V, Villa-Gonzalez E, Aguilar-Farias N, Rodriguez-Rodriguez F. Reliability, reproducibility, and feasibility of youth activity profile (YAP) questionnaire in Chilean children and adolescents. J Sports Sci. 2024 Oct;42(20):1959-1966. doi: 10.1080/02640414.2024.2419278. Epub 2024 Oct 24. PMID 39445725
- [Background] Saint-Maurice PF, Welk GJ. Validity and Calibration of the Youth Activity Profile. PLoS One. 2015 Dec 2;10(12):e0143949. doi: 10.1371/journal.pone.0143949. eCollection 2015. PMID 26630346
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Tremblay MS, Carson V, Chaput JP. Introduction to the Canadian 24-Hour Movement Guidelines for Children and Youth: An Integration of Physical Activity, Sedentary Behaviour, and Sleep. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):iii-iv. doi: 10.1139/apnm-2016-0203. No abstract available. PMID 27306430
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350